CLINICAL TRIAL: NCT02697253
Title: Mechanisms Underlying Predictors of Success From Obesity Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Harry Kissileff, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GCO 15-1990; R01DK108643 (NIH); AAAQ1904 (Other: Columbia University Medical Center)
Record Dates: First submitted 2016-02-23; First posted 2016-03-03 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Obesity
Keywords: Roux-en-Y Bariatric Surgery; Psychosocial Variables; Behavioral Variables; Weight Loss; Food Intake; GLP-1; Reinforcing Value of Food; Exendin 9-39
MeSH Terms: conditions — Obesity; Weight Loss | interventions — exendin (9-39); Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Successful drug (Experimental): Participants who have a % weight loss ≥35 at 2 years post RYGB/SG surgery will be administered sitagliptin and receive infusion of Exendin 9-39 prior to an intake test.
  Drug: Exendin 9-39 Infusion of exendin 9-39 at the rate of 600 pmol/kg/min, infusion time 80 minutes. An average of 18.2mg will be infused in a forearm vein during an oral glucose (30g) preload.
  Drug: Sitagliptin 100mg tablet will be administered at 2200 hours the night before the visit. The day of the visit, the patient will take another 100mg tablet at 0700 hours.
  Interventions: Drug: Exendin 9-39 and Sitagliptin
- Unsuccessful drug (Experimental): Participants who have a % weight loss of ≤25 at two years post RYGB/SG surgery will be administered Sitagliptin and receive infusion of Exendin 9-39 prior to an intake test.
  Drug: Exendin 9-39 Infusion of exendin 9-39 at the rate of 600 pmol/kg/min, infusion time 80 minutes. An average of 18.2mg will be infused in a forearm vein during an oral glucose (30g) preload.
  Drug: Sitagliptin 100mg tablet will be administered at 2200 hours the night before the visit. The day of the visit, the patient will take another 100mg tablet at 0700 hours.
  Interventions: Drug: Exendin 9-39 and Sitagliptin
- Success placebo (Placebo Comparator): Participants who have a % weight loss ≥35 at 2 years post RYGB/SG surgery will be administered a placebo and receive a placebo infusion prior to an intake test.
  Drug: Placebo Infusion of 0.9% saline solution (placebo infusion) for 80 minutes. An average of 18.2mg will be infused in a forearm vein during an oral glucose (30g) preload.
  Drug: Placebo 100mg tablet will be administered at 2200 hours the night before the visit. The day of the visit, the patient will take another 100mg tablet at 0700 hours.
  Interventions: Drug: Placebo
- Unsuccess placebo (Placebo Comparator): Participants who have a % weight loss of ≤25 at two years post RYGB/SG surgery will be administered a placebo and receive a placebo infusion prior to an intake test.
  Drug: Placebo Infusion of 0.9% saline solution (placebo infusion) for 80 minutes. An average of 18.2mg will be infused in a forearm vein during an oral glucose (30g) preload.
  Drug: Placebo 100mg tablet will be administered at 2200 hours the night before the visit. The day of the visit, the patient will take another 100mg tablet at 0700 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exendin 9-39 and Sitagliptin — Infusion of exendin 9-39 at the rate of 600 pmol/kg/min, infusion time 80 minutes. An average of 18.2mg will be infused in a forearm vein during an oral glucose (30g) preload.
  100mg tablet will be administered at 2200 hours the night before the visit. The day of the visit, the patient will take another 100mg tablet at 0700 hours.
  Arms: Successful drug; Unsuccessful drug
Drug: Placebo — Infusion of 0.9% saline solution (placebo infusion) for 80 minutes. An average of 18.2mg will be infused in a forearm vein during an oral glucose (30g) preload.
  100mg Placebo tablet will be administered at 2200 hours the night before the visit. The day of the visit, the patient will take another 100mg placebo tablet at 0700 hours.
  Arms: Success placebo; Unsuccess placebo

SUMMARY:
The goal of this project is to identify predictors of success in the treatment of obesity after bariatric surgery. The specific aims of this proposal are to:

1. Employ behavioral tests of mechanisms that control food intake in normal weight individuals, to determine which intake control mechanisms lead to changes after Roux-en-y gastric bypass (RYGB) or sleeve gastrectomy (SG); and
2. Measure behavioral and psycho-social predictors of weight loss and food intake reduction, so as to determine which are most predictive of successful weight loss and food intake reduction.
3. Account for success in reduction of food intake brought about by the pattern of hormone release, particularly glucagon-like peptide-1 (GLP-1), Peptide YY (PYY) and gastric distention, known to underlie satiation, coupled with post-ingestive changes in reinforcing value of food and motivation to consume.

Tests of the hypothesis will be done by measuring responses to tasting, working for, and consuming, foods on sensory, motivational, cognitive, and physiological variables, including amount consumed and rate of eating under standardized conditions, before surgery and at a two year follow up visit. In addition, the inhibitor sitagliptin will be administered the night before and day of test meal and exendin-9-39 (EX9) will be infused before and during the meal to determine whether blockade of GLP-1 / PYY receptors after surgery reverses intake reduction. Investigators predict that successful patients will show changes that favor reduction in food intake, rate of eating, motivation to consume, reward value of foods, and a hormone profile that has been shown to generate satiation and maintain reduction in intake (e.g. increased Cholecystokinin (CCK), GLP-1, PYY, reduced ghrelin). To the extent that psycho-social and cognitive factors may override physiological brakes to eating behavior, the subjects may fail to achieve success, and consequently the failure may be predicted from over-impulsiveness or inability to suppress working for rewarding food stimuli. To test these hypotheses, a total of 83 patients will be enrolled prior to RYGB/SG and restudied 2 years after the surgery. The sitagliptin / EX9 studies will be done in a subset of 32 completers. To test this aim, patients will be divided into 4 groups of 19. The 4 patients from each group with the most weight loss (% weight loss ≥35 at 2 years post-surgery, 16 patients in total) and least weight loss (% weight loss of ≤25 at two years 16 patients in total) will be recruited for these two additional post-operative visits within one year of completing Visit #3 after the RYGB/SG surgery. A total of 32 patients will be recruited for visits 4 and 5.

DETAILED DESCRIPTION:
Obesity is a major public health as well as economic (expense of treating) problem world-wide, and Roux-en-Y gastric bypass (RYGB) and Sleeve Gastrectomy (SG) surgeries are effective treatments. A barrier to progress is that between 25% and 40% patients were not successful in achieving and maintaining at least 30% weight loss, which is considered medically successful for this operation. Understanding the mechanisms that contribute to success or failure of this operation is an unsolved problem in obesity research, which this proposal is addressing. The focus of this project is to identify mechanisms that contribute to suppression of food intake following bariatric surgery, and to investigate whether these mechanisms predict long-term success following bariatric surgery

ELIGIBILITY:
Inclusion Criteria:

* BMI >35 kg/m2 BMI
* BMI < 65 kg/m2
* Preparing to undergo Roux-en-Y gastric bypass or gastric sleeve (RYGB/GS) surgery at St. Luke-Roosevelt Hospital
* Within the 18-65 age range
* Blood pressure under <160/100 mmHg
* Fasting triglyceride <600 mg/dl
* No recent (last 6 months) history of cardiovascular disease.
* Prior history of angioplasty or coronary artery bypass surgery with a normal stress test will not be a contraindication.

Exclusion Criteria:

* Diabetes Mellitus
* Active cancer
* Unstable angina
* Recent stroke
* Current therapy that may affect glucose metabolism such as glucocorticoids, adrenergic agents
* Active infection
* Kidney failure
* Severe liver dysfunction
* Heavy alcohol use
* Severe respiratory or cardiac failure
* Pancreatitis
* History of bullous pemphigoid
* Pregnancy
* Patients who are currently or have had prior GLP-1 therapy.
* Patients with known hypersensitivity to Exendin 9-39 or similar products, albumin, sitagliptin and/or acetaminophen will also be excluded.

Additional exclusions for visits 4 and 5 ONLY:

* Patients at risk for heart disease, such as patients with a history of atherosclerotic cardiovascular disease and history of heart failure
* Renal impairment (eGFR˂60 Ml/MIN/1.73 M2)
* History of exfoliative skin conditions in particularly if occurring with a DPP-4 inhibitor use
* History of bullous pemphigoid and Stevens-Johnson syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Successful Weight Loss | 2 years
  % Excess body weight lost

SECONDARY OUTCOMES:
Intake amount in grams consumed in a food intake capacity test | 2 years
  Intake amount in grams consumed in a food intake capacity test
Fullness levels based on a rating scale after food intake capacity test | 2 years
  Fullness levels based on a rating scale after food intake capacity test
Sickness levels based on a rating scale after food intake capacity test | 2 years
  Sickness levels based on a rating scale after food intake capacity test

CONTACTS AND LOCATIONS:
Overall Officials: Harry Kissileff, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai - Morningside, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No